CLINICAL TRIAL: NCT06079125
Title: Type of Surgical Intervention for Chiari Malformation-syringomyelia: a Multicenter Randomized Controlled Study
Brief Title: PFDD Versus PFDRT in Chiari Decompression Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DDCS
Record Dates: First submitted 2023-08-20; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Chiari Malformation Type I; Tonsillectomy
Keywords: posterior fossa decompression with duraplasty; tonsillectomy; FMDD
MeSH Terms: conditions — Arnold-Chiari Malformation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posterior fossa decompression with duraplasty (Experimental): The bone is removed from the suboccipital region of the skull and Cervical 1 lamina so the constricting epidural band can be resected. Then, the dura is opened. Microsurgical dissection is performed and the dura is sewn closed.
  Interventions: Procedure: Posterior fossa decompression with duraplasty
- PFDD with tonsillar resection/reduction (Experimental): The bone is removed from the suboccipital region of the skull and Cervical 1 lamina so the constricting epidural band can be resected. Then, the dura is opened and herniated tonsil will be manipulated. Microsurgical dissection is performed and the dura is sewn closed.
  Interventions: Procedure: PFDD with tonsillar resection/reduction

INTERVENTIONS:
Procedure: Posterior fossa decompression with duraplasty — The dura is opened sharply, exposing the cerebellar tonsils, brainstem, and upper spinal cord. After microsurgical dissection, the dura is sewn closed with a dural graft.
  Arms: Posterior fossa decompression with duraplasty
Procedure: PFDD with tonsillar resection/reduction — The dura is opened sharply, exposing the cerebellar tonsils, brainstem, and upper spinal cord. Then herniated tonsil will be manipulated and adhesion was released. After microsurgical manipulated, the dura is sewn closed with a dural graft.
  Arms: PFDD with tonsillar resection/reduction

SUMMARY:
The purpose of this study is to determine whether a posterior fossa decompression and duraplasty with or without tonsil manipulation results in better patient outcomes with fewer complications and improved quality of life in those who have Chiari malformation type I and syringomyelia.

DETAILED DESCRIPTION:
Participants with Chiari Malformation type I and syringomyelia will be randomized to either have a posterior fossa decompression and duraplasty with or without tonsil manipulation. The participant will then return to the neurosurgeon's office at the following time points which are consistent with standard of care practice: 3-6 months, 12 and 24 months. At these visits, the clinician will complete a physical exam and the participant will report on the prognosis of symptoms and complete questionnaires. A spine MRI will be performed 3-6 months, 12 and 24 months after the decompression.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥14 years old
* Chiari malformation type I ≥5 mm tonsillar ectopia
* a syrinx with a width > 50% of the cross-sectional diameter of the spinal cord , and a length of at least 2 cervical and/or thoracic vertebral segments.
* MRI of the brain and cervical and thoracic spine are required prior to surgery and must be available to be shared with the Data Coordinating Center

Exclusion Criteria:

* included one or more of the following preexisting conditions: hydrocephalus; tumor; brain trauma; stroke; meningitis; abscess;
* other congenital anomalies of the brain or skull base; vertebral anomalies (i.e., Klippel-Feil, atlas assimilation, etc.);
* degenerative or demyelinating disease;
* CM-I without syringomyelia;
* syringomyelia with cerebellar tonsils in a normal position;
* fibromyalgia;
* chronic fatigue syndrome;
* prior posterior fossa surgery.
* Unable to share pre-decompression MRI of the brain and spine Patients who do not wish to participate

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
improvement or resolution of the syrinx, | 3-6, 12 and 24 months
  defined as > 50% improvement in length, maximal cross-sectional diameter, or both.

SECONDARY OUTCOMES:
complication rates | 12 months
  Reoperation,Wound infection,Aseptic meningitis,CSF fistula,Subcutaneous hydrops,Other complications
Chicago Chiari Outcome Scale (CCOS) scale | 12 months
visual analog scale (VAS) | 12 months
  degree of the pain
Japanese Orthopaedic Association (JOA) scale | 12 months
  Japanese Orthopaedic Association Scores
blood loss | 12 months
  blood loss
hospital stay | 12 months
  hospital stay
cost for the hospitalisation. | 12 months
  cost for the hospitalisation.

CONTACTS AND LOCATIONS:
Overall Officials: fengzeng jian, Study Chair — Xuanwu Hospital, Beijing
Locations (1):
- Fengzeng Jian, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hale AT, Adelson PD, Albert GW, Aldana PR, Alden TD, Anderson RCE, Bauer DF, Bonfield CM, Brockmeyer DL, Chern JJ, Couture DE, Daniels DJ, Durham SR, Ellenbogen RG, Eskandari R, George TM, Grant GA, Graupman PC, Greene S, Greenfield JP, Gross NL, Guillaume DJ, Heuer GG, Iantosca M, Iskandar BJ, Jackson EM, Johnston JM, Keating RF, Leonard JR, Maher CO, Mangano FT, McComb JG, Meehan T, Menezes AH, O'Neill B, Olavarria G, Park TS, Ragheb J, Selden NR, Shah MN, Smyth MD, Stone SSD, Strahle JM, Wait SD, Wellons JC, Whitehead WE, Shannon CN, Limbrick DD; Park-Reeves Syringomyelia Research Consortium Investigators. Factors associated with syrinx size in pediatric patients treated for Chiari malformation type I and syringomyelia: a study from the Park-Reeves Syringomyelia Research Consortium. J Neurosurg Pediatr. 2020 Mar 6;25(6):629-639. doi: 10.3171/2020.1.PEDS19493. Print 2020 Jun 1. PMID 32114543
- [Background] Yuan C, Wei M, Li W, Wang X, Jian F. Comparison of Foramen Magnum Decompression with and without Duraplasty in the Treatment of Adult Chiari Malformation Type I: A Meta-Analysis and Systematic Review. Turk Neurosurg. 2022;32(6):893-902. doi: 10.5137/1019-5149.JTN.35727-21.5. PMID 35652180
- [Background] Guan J, Yuan C, Zhang C, Ma L, Yao Q, Cheng L, Liu Z, Wang K, Duan W, Wang X, Wu H, Chen Z, Jian F. Intradural Pathology Causing Cerebrospinal Fluid Obstruction in Syringomyelia and Effectiveness of Foramen Magnum and Foramen of Magendie Dredging Treatment. World Neurosurg. 2020 Dec;144:e178-e188. doi: 10.1016/j.wneu.2020.08.068. Epub 2020 Aug 15. PMID 32805463
- [Background] Yuan C, Guan J, Du Y, Zhang C, Ma L, Yao Q, Cheng L, Liu Z, Wang K, Duan W, Wang X, Wu H, Chen Z, Jian F. Repeat Craniocervical Decompression in Patients with a Persistent or Worsening Syrinx: A Preliminary Report and Early Results. World Neurosurg. 2020 Jun;138:e95-e105. doi: 10.1016/j.wneu.2020.02.015. Epub 2020 Feb 12. PMID 32059967
- [Background] Heiss JD, Jarvis K, Smith RK, Eskioglu E, Gierthmuehlen M, Patronas NJ, Butman JA, Argersinger DP, Lonser RR, Oldfield EH. Origin of Syrinx Fluid in Syringomyelia: A Physiological Study. Neurosurgery. 2019 Feb 1;84(2):457-468. doi: 10.1093/neuros/nyy072. PMID 29618081
- [Background] Koueik J, Sandoval-Garcia C, Kestle JRW, Rocque BG, Frim DM, Grant GA, Keating RF, Muh CR, Oakes WJ, Pollack IF, Selden NR, Tubbs RS, Tuite GF, Warf B, Rajamanickam V, Broman AT, Haughton V, Rebsamen S, George TM, Iskandar BJ. Outcomes in children undergoing posterior fossa decompression and duraplasty with and without tonsillar reduction for Chiari malformation type I and syringomyelia: a pilot prospective multicenter cohort study. J Neurosurg Pediatr. 2019 Oct 18;25(1):21-29. doi: 10.3171/2019.8.PEDS19154. Print 2020 Jan 1. PMID 31628281